CLINICAL TRIAL: NCT02238405
Title: A Randomized Controlled Smoking Cessation Trial and Prospective Cohort Study of TB Treatment Outcomes
Brief Title: A Controlled Smoking Cessation Trial and Prospective Cohort Study of Tuberculosis (TB) Treatment Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Global Fund (Other); National Tuberculosis Control Program, Pakistan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00037636
Record Dates: First submitted 2014-07-22; First posted 2014-09-12 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Smoking Cessation; Tuberculosis
MeSH Terms: conditions — Smoking Cessation; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counseling (Experimental): Intensive anti-smoking counseling
  Interventions: Other: Intensive anti-smoking counseling
- Standard Care (No Intervention): Control group will receive current standard of care.

INTERVENTIONS:
Other: Intensive anti-smoking counseling — Study participants randomized to the intervention arm will receive intensive cessation support outside of the TB clinic setting, from a health worker trained in cessation counseling, during the course of their TB treatment. Behavioral elements will consist of follow up using unscheduled drop in or phone sessions, motivational interviewing, and counseling tailored to the needs and circumstances of the patient. Patients who are current smokers and are ready to commit to quit smoking will be supported to stop completely. Recent smokers will supported for having quit, and the counselor will discuss coping strategies to maintain abstinence.
  Arms: Counseling

SUMMARY:
The primary focus of this intervention trial is to understand the effect of quitting smoking on TB treatment outcomes. The investigators will compare a cessation strategy based on guidelines recommended by the World Health Organization (WHO) and the International Union against Tuberculosis and Lung Disease (IUTLD). This is currently not utilized in TB directly observed therapy (DOT) clinics in Pakistan. The investigators study will provide comprehensive data towards understanding the effectiveness of these strategies for TB patients who smoke in Pakistan, and most importantly, on the effect of quitting smoking on TB treatment outcomes. These findings will guide development of effective smoking cessation strategies in a region with high prevalence of TB and increasing tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* Males, ≥18 years of age
* diagnosed with pulmonary TB
* self-reported current smokers, or smoker within 6 months
* anticipated to be attending the TB treatment clinic for at least 6 months
* be willing to set a quit date within 2 weeks after baseline assessment
* agree to participate

Exclusion Criteria:

* less than 18 years of age
* quit for more than 6 months
* extra-pulmonary TB
* unable/unwilling to provide written consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2015-05-25 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Smoking cessation rate | 1-6 months
Smoking cessation rate | 6 months post-TB treatment

SECONDARY OUTCOMES:
negative TB treatment outcome (death, treatment failure, relapse, required prolongation of TB therapy | 6 months post-TB treatment
  To assess differences in TB treatment outcomes between smokers and quitters, all patients enrolled in the intervention trial will be included in analyses of a composite negative outcome variable, defined as a composite endpoint of poor clinical response to TB treatment including death, treatment failure, relapse, and/or requirement for prolongation of TB therapy. Risk of a negative treatment outcome will be compared between the following 3 groups: 1) TB patients who were current smokers and quit smoking for 6 months of follow-up; 2) TB patients who were recent smokers and stayed quit for 6 months of follow-up; and, 3) TB patients who are never smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan E Golub, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Indus Hospital, Karachi, Pakistan